CLINICAL TRIAL: NCT01065909
Title: National Observatory on the Therapeutic Management in Ambulatory Care Patients Aged 65 and Over, With Diabetes Type 2, Chronic Pain or Atrial Fibrillation
Brief Title: Observatory on Elderly Patients "Les S.AGES"
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: DIREG_L_04182
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Pain; Atrial Fibrillation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Pain; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Diabetes type 2
- Chronic Pain
- Atrial Fibrillation

SUMMARY:
Primary objective shared by the 3 registries : Describe the different pharmacotherapeutic management in patients :

* DB (Diabetes): with type 2 diabetes, treated with oral and / or injectable antidiabetics
* CP (Chronic Pain): with any disease leading to chronic pain (lasting for more than 3 months)
* AF (Atrial Fibrillation): with ongoing AF or AF diagnosed within 12 months before enrollment

Secondary objectives shared by the 3 observatories:

* Describe the occurrence of clinical events, hospitalizations and death, according to the different medical care conditions, and analyze their predicting factors
* Estimate the resources consumption according to the medical and non medical management of these patients,
* Analyze the impact of some factors (patient's cognitive status, autonomy, renal function ...) on the current practice

Secondary objectives specific shared by DB and AF registries :

- Analyze the geriatric pharmaco-genetic aspects

Specific secondary objectives for each observatory :

* DB : Describe HbA1c level, percentage of responders and body weight evolution according to the different medical care conditions
* CP : Evaluate pain consequences on Daily Living Activities and patient autonomy

ELIGIBILITY:
Inclusion Criteria specific for each observatory :

* DB : Established type 2 diabetes treated with oral and / or injectable antidiabetics
* CP : Pain lasting for over 3 months, requiring therapeutic care
* FA : Ongoing Atrial fibrillation or AF diagnosed within the 12 months before enrollment and documented by ECG or Holter ECG, whatever the rhythm at inclusion

Exclusion Criteria shared by the 3 observatories:

* Living in accommodation facility for dependent patients
* Patient with non cardiovascular progressively unstable disease
* Patient already enrolled in a clinical trial
* Patient unlikely to complete the study

Exclusion Criteria specific for just AF observatory :

- Transitional AF due to thyrotoxicosis, alcohol, myocarditis, pericarditis, acute myocardial infarction, pulmonary embolism, metabolic disorders or electrocution, Post cardiac surgery AF (<3 months).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Ambulatory primary care patient over 65 years
Sampling Method: Non-Probability Sample
Enrollment: 3491 (Actual)
Dates: Start 2009-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France

REFERENCES:
- [Derived] Strumia M, Vidal JS, Cestac P, Sallerin B, Andrieu S, Hanon O, Rouch L; S.AGES investigators *. Blood Pressure Postural Changes Variability Is Associated With Lower Cognition: The S.AGES Cohort. J Am Heart Assoc. 2025 Oct 7;14(19):e039197. doi: 10.1161/JAHA.124.039197. Epub 2025 Oct 8. PMID 41059541
- [Derived] Baudouin E, Colle R, Becquemont L, Corruble E, Duron E. Association between driving and depression in older adults: findings from an ancillary study of a prospective cohort. BMC Geriatr. 2025 Mar 14;25(1):173. doi: 10.1186/s12877-025-05826-8. PMID 40087594
- [Derived] Zitoun S, Baudouin E, Corruble E, Vidal JS, Becquemont L, Duron E. Use of potentially driver-impairing drugs among older drivers. BMC Geriatr. 2022 Jan 3;22(1):4. doi: 10.1186/s12877-021-02726-5. PMID 34979970
- [Derived] Hanon O, Vidal JS, Pisica-Donose G, Benattar-Zibi L, Bertin P, Berrut G, Corruble E, Derumeaux G, Falissard B, Forette F, Pasquier F, Pinget M, Ourabah R, Becquemont L, Danchin N; S.AGES Investigators. Therapeutic management in ambulatory elderly patients with atrial fibrillation: the S.AGES cohort. J Nutr Health Aging. 2015 Feb;19(2):219-27. doi: 10.1007/s12603-015-0444-9. PMID 25651449
- [Derived] Bucher S, Bauduceau B, Benattar-Zibi L, Bertin P, Berrut G, Corruble E, Danchin N, Delespierre T, Derumeaux G, Doucet J, Falissard B, Forette F, Hanon O, Ourabah R, Pasquier F, Piedvache C, Pinget M, Ringa V, Becquemont L; S.AGES Investigators. Primary care management of non-institutionalized elderly diabetic patients: The S.AGES cohort - Baseline data. Prim Care Diabetes. 2015 Aug;9(4):267-74. doi: 10.1016/j.pcd.2014.07.004. Epub 2014 Jul 31. PMID 25086913
- [Derived] Bertin P, Becquemont L, Corruble E, Derumeaux G, Falissard B, Hanon O, Pinget M, Forette F. The therapeutic management of chronic pain in ambulatory care patients aged 65 and over in France: the S.AGES Cohort. Baseline data. J Nutr Health Aging. 2013;17(8):681-6. doi: 10.1007/s12603-013-0338-7. PMID 24097022